CLINICAL TRIAL: NCT04401098
Title: Survey Of Egyptian Population Change in Knowledge, Attitude and Behaviour Towards COVID 19 Outbreak
Brief Title: Changing Of Egyptian Population Behaviour Towards COVID 19 Outbreak
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Damanhour University (Other)
Responsible Party: Sponsor
Other Study IDs: covid 19
Record Dates: First submitted 2020-05-22; First posted 2020-05-26 (Actual); Last update posted 2020-05-26 (Actual); Status verified 2020-05

CONDITIONS: COVID 19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
During the COVID-19 pandemic, the Egyptian government issued movement restrictions and placed areas into quarantine to reduce the spread of the disease. In addition, individuals were encouraged to adopt personal protective measures, such as social isolation , increasing personal hygiene and wearing protective face masks. Information regarding the COVID 19 virus and protective measures is found on social media and ministry of health website and a number of the Egyptian population are keeping track of them .Public Awareness play a major rule in reducing the spread of COVID 19 so in this study a survey is done to measure the awareness of the Egyptian population toward COVID 19 , their knowledge and attitude and their adherence to preventive measures.It also measures the change of their behavior during the beginning of the outbreak and after a few months of the outbreak in Egypt.

DETAILED DESCRIPTION:
Detailed Description:

The survey will enroll as many individuals of the Egyptian population as possible in the survey portion of the study - The number of participates have no limitations, at least 700 participants.

The survey will be enrolled in online google form, face to face interview(this will be reduced to encourage social isolation) & semi-structured telephone interviews if possible.

The research procedures:

An online survey link will include questions regarding the awareness of the Egyptian population , their knowledge , attitudes and behaviour during covid-19 outbreak.and also a comparison of their behaviour among different time periods of the outbreak Face to face and semi-structured interviews if possible: For those Egyptian citizens who state that they would like to participate in an interview, a random sample will be contacted.

Inclusion Criteria:

Egyptian population of any age group

Exclusion Criteria:

none

ELIGIBILITY:
Inclusion Criteria:

Egyptian population of different age groups

Exclusion Criteria:

none

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: any individual of the Egyptian population of any age group.
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2020-05-02 (Actual); Primary Completion 2020-10-01 (Estimated); Study Completion 2021-04-01 (Estimated)

PRIMARY OUTCOMES:
awareness of Egyptian population | 6 months
  evaluate the knowledge , attitude and behaviour and their change among Egyptian population during COVID 19 outbreak.

CONTACTS AND LOCATIONS:
Locations (1):
- Damanhour University, Damanhur, Beheira, Egypt

IPD SHARING:
Plan to Share IPD: Undecided